CLINICAL TRIAL: NCT05032183
Title: Phase Ib/II Study of the Combination of Low-Intensity Chemotherapy and Tagraxofusp in Patients With Acute Lymphoblastic Leukemia (ALL)
Brief Title: Tagraxofusp and Low-Intensity Chemotherapy for the Treatment of CD123 Positive Relapsed or Refractory Acute Lymphoblastic Leukemia or Lymphoblastic Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to slow enrollment.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0545; NCI-2021-08859 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0545 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-23; First posted 2021-09-02 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Adult Lymphoblastic Lymphoma; Recurrent B Acute Lymphoblastic Leukemia; Recurrent T Acute Lymphoblastic Leukemia; Refractory B Acute Lymphoblastic Leukemia; Refractory Lymphoblastic Lymphoma; Refractory T Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; Cytarabine; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Filgrastim; Granulocyte Colony-Stimulating Factor; Leucovorin; Mercaptopurine; azathiopurine; Mesna; Methotrexate; merphos; pegfilgrastim; Prednisone; deltacortene; prednylidene; Rituximab; CT-P10; tagraxofusp; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (tagraxofusp, chemotherapy) (Experimental): See Detailed Description
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Biological: Filgrastim-sndz; Drug: Leucovorin; Drug: Mercaptopurine; Drug: Mesna; Drug: Methotrexate; Biological: Pegfilgrastim; Drug: Prednisone; Biological: Rituximab; Biological: Tagraxofusp-erzs; Drug: Vincristine

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IT
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Biological: Filgrastim-sndz — Given SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Zarxio
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Mesna — Give IV
  Other Names: 2-Mercaptoethanesulfonate, Sodium Salt; Ausobronc; D-7093; Filesna; Mercaptoethane Sulfonate; Mercaptoethanesulfonate; Mesnex; Mesnil; Mesnum; Mexan; Mistabron; Mistabronco; Mitexan; Mucofluid; Mucolene; UCB 3983; Uromitexan; Ziken
Drug: Methotrexate — Given IT
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Biological: Pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; filgrastim-SD/01; Fulphila; HSP-130; Jinyouli; Neulasta; Neulastim; Nyvepria; Pegcyte; Pegfilgrastim Biosimilar HSP-130; Pegfilgrastim Biosimilar Nyvepria; Pegfilgrastim Biosimilar Pegcyte; Pegfilgrastim Biosimilar Udenyca; Pegfilgrastim Biosimilar Ziextenzo; pegfilgrastim-apgf; pegfilgrastim-bmez; pegfilgrastim-cbqv; Pegfilgrastim-jmdb; SD-01; SD-01 sustained duration G-CSF; Udenyca; Ziextenzo
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima
Biological: Tagraxofusp-erzs — Given IV
  Other Names: Diphtheria Toxin(388)-Interleukin-3 Fusion Protein; DT(388)-IL3 Fusion Protein; DT388IL3 fusion protein; Elzonris; IL3R-targeting Fusion Protein SL-401; SL-401; Tagraxofusp; Tagraxofusp ERZS
Drug: Vincristine — Given IV
  Other Names: Leurocristine; VCR; Vincrystine

SUMMARY:
This phase Ib/II trial studies the effects of tagraxofusp and low-intensity chemotherapy in treating patients with CD123 positive acute lymphoblastic leukemia or lymphoblastic lymphoma that has come back (relapsed) or does not respond to treatment (refractory). Tagraxofusp consists of human interleukin 3 (IL3) linked to a toxic agent called DT388. IL3 attaches to IL3 receptor positive cancer cells in a targeted way and delivers DT388 to kill them. Chemotherapy drugs, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving tagraxofusp with chemotherapy may help control CD123 positive relapsed or refractory acute lymphoblastic leukemia or lymphoblastic lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the overall response rate (complete response [CR] + CR with inadequate count recovery [CRi]) of the regimen within 3 cycles.

SECONDARY OBJECTIVES:

I. Evaluate other clinical efficacy endpoints (CR rate, minimal residual disease [MRD] negativity, duration of response [DOR], relapse-free survival [RFS] overall survival [OS]).

II. Determine the proportion of patients proceeding to allogeneic stem cell transplantation (allo-SCT).

III. Determine the safety of the combination regimen.

EXPLORATORY OBJECTIVES:

I. To determine CD123 expression levels pre- and post-therapy. II. To correlate baseline CD123 expression with response rates and duration of response.

III. To evaluate change in apoptotic protein expression and alterations in cellular signaling pathways using cytometry by time of flight (CyTOF).

IV. To determine baseline gene expression profile in order to identify ALL subtypes and correlate with clinical outcomes and response to single-agent tagraxofusp-erzs (tagraxofusp).

OUTLINE:

TAGRAXOFUSP AND CHEMOTHERAPY PHASE:

CYCLE 1: Patients receive tagraxofusp-erzs intravenously (IV) over 15 minutes on days 1-5.

CYCLES 2 AND 4: Patients receive tagraxofusp-erzs IV over 15 minutes on days 1-3, cyclophosphamide IV over 3 hours twice daily (BID) and mesna IV on days 4-6, vincristine IV over 15 minutes on days 4 and 15, dexamethasone IV over 30 minutes or orally (PO) on day 4-7 and 14-17, methotrexate intrathecally (IT) on day 5, and filgrastim-sndz subcutaneously (SC) or pegfilgrastim SC on day 8, and cytarabine IT on day 10. Patients may receive rituximab IV over 4-6 hours on days 4 and 14.

CYCLES 3 AND 5: Patients receive tagraxofusp-erzs IV over 15 minutes on days 1-3, methotrexate IV over 24 hours on day 4, cytarabine IV over 3 hours BID on days 5-6, filgrastim-sndz SC or pegfilgrastim SC on day 6, methotrexate IT and cytarabine IT on day 11. Patients may receive rituximab IV over 4-6 hours on days 4 and 11. Beginning about 12 hours after the day 4 dose of methotrexate, patients may also receive leucovorin IV over 15 minutes, 4 times a day for about 8 doses.

CYCLES 6 AND 8: Patients receive cyclophosphamide IV over 3 hours BID and mesna IV on days 1-3, vincristine IV over 15 minutes on days 1 and 11, dexamethasone IV over 30 minutes or PO on day 1-4 and 11-14, and filgrastim-sndz SC or pegfilgrastim SC on day 5.

CYCLES 7 AND 9: Patients receive methotrexate IV over 24 hours on day 1, cytarabine IV over 3 hours BID on days 2-3, and filgrastim-sndz SC or pegfilgrastim SC on day 4. Beginning about 12 hours after the day 1 dose of methotrexate, patients may receive leucovorin IV over 15 minutes, 4 times a day for about 8 doses.

Cycle 1 is 21 days. Treatment repeats every 28 days for cycles 2-9 in the absence of disease progression or unacceptable toxicity.

TAGRAXOFUSP AND MAINTENANCE PHASE:

CYCLES 1-3, 5-7, 9-11, 13-15: Patients receive mercaptopurine PO three time daily (TID) on days 1-28, prednisone PO once daily (QD) on day 1-5, methotrexate PO once every week (QW) and vincristine IV over 15 minutes every 4 weeks.

CYCLES 4, 8, and 12: Patients receive tagraxofusp-erzs IV over 15 minutes on days 1-5.

Treatment repeats every 28 days for 15 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-70 years of age with relapsed/refractory CD123+ B- or T-cell acute lymphoblastic leukemia (ALL) or lymphoblastic lymphoma. CD123 positivity may be confirmed by either flow cytometry or immunohistochemistry
* Performance status =< 2 (Eastern Cooperative Oncology Group [ECOG] scale)
* Total serum bilirubin =< 1.5 x upper limit of normal (ULN), unless due to Gilbert's syndrome, in which case patients are eligible as long as direct bilirubin =< 2 x ULN
* Alanine aminotransferase (ALT) =< 2.5 x ULN, unless due to disease involvement of the liver or hemolysis, in which case an ALT =< 10 x ULN is acceptable
* Aspartate aminotransferase (AST) =< 2.5 x ULN, unless due to disease involvement of the liver or hemolysis, in which case an ALT =< 10 x ULN is acceptable
* Serum creatinine =< 1.5 mg/dL
* Serum albumin >= 3.2 g/dL (32 g/L). Albumin infusions are not permitted in order to enable eligibility
* For females of childbearing potential, a negative pregnancy test must be documented within 1 week of starting treatment
* Female and male patients who are fertile must agree to use an effective form of contraception (birth control methods while on study, such as birth control pills or injections, intrauterine devices (IUDs), or double-barrier methods (for example, a condom in combination with spermicide) with their sexual partners for 4 months after the end of treatment
* Signed informed consent
* Willingness and ability to adhere to study visit schedule and other protocol requirements, including follow-up for survival assessment

Exclusion Criteria:

* Active serious infection not controlled by oral or intravenous antibiotics
* Known active central nervous system (CNS) leukemia
* Diagnosis of Philadelphia chromosome-positive ALL or Burkitt leukemia/lymphoma
* Active graft versus host disease (GVHD)
* Active secondary malignancy other than skin cancer (e.g., basal cell carcinoma or squamous cell carcinoma) that in the investigator's opinion will shorten survival to less than 1 year
* Known hepatitis B or C infection, or known seropositivity for human immunodeficiency virus (HIV)
* Clinically significant cardiovascular disease (e.g., uncontrolled or any New York Heart Association Class 3 or 4 congestive heart failure, uncontrolled angina, history of myocardial infarction, unstable angina or stroke within 6 months prior to study entry, uncontrolled hypertension or clinically significant arrhythmias not controlled by medication)
* Patients with a cardiac ejection fraction (as measured by either multigated acquisition [MUGA] or echocardiogram) less than the lower limit of normal
* No clinically significant abnormalities on 12-lead electrocardiogram
* Uncontrolled, clinically significant pulmonary disease (e.g., chronic obstructive pulmonary disease, pulmonary hypertension) that in the opinion of the Investigator would put the patient at significant risk for pulmonary complications during the study
* Persistent clinically significant toxicities grade >= 2 from previous chemotherapy (excluding alopecia, nausea, fatigue, and liver function tests [as mandated in the inclusion criteria])
* Treatment with any investigational antileukemic agents or chemotherapy agents in the last 7 days before study entry, unless full recovery from side effects has occurred or patient has rapidly progressive disease judged to be life-threatening by the investigator. Exception: Treatment with hydroxyurea and/or dexamethasone are allowed prior to study treatment, without window of exclusion
* Pregnant and lactating women will not be eligible; women of childbearing potential should have a negative pregnancy test prior to entering on the study and be willing to practice methods of contraception for 4 months after last study treatment. Women do not have childbearing potential if they have had a hysterectomy or are postmenopausal without menses for 12 months. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control for 4 months after last study treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Short, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Treatment (Tagraxofusp, Chemotherapy): See Detailed Description
  Cyclophosphamide: Given IV
  Cytarabine: Given IT
  Dexamethasone: Given IV or PO
  Filgrastim-sndz: Given SC
  Leucovorin: Given IV
  Mercaptopurine: Given PO
  Mesna: Give IV
  Methotrexate: Given IT
  Pegfilgrastim: Given SC
  Prednisone: Given PO
  Rituximab: Given IV
  Tagraxofusp-erzs: Given IV
Period: Overall Study
Arm/Group | Phase I Treatment (Tagraxofusp, Chemotherapy)
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phase I Treatment (Tagraxofusp, Chemotherapy)
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Age, Continuous [Median (Full Range); unit: Years] | 31 [19 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Response
Description: Response is defined as Complete Response CR + Complete Response with inadequate count recovery (CRi) - (CR): Normalization of the peripheral blood and bone marrow with 5% or less blasts in normocellular or hypercellular marrow with a granulocyte count of 1 x 10^9/L or above, and platelet count of 100 x 10^9/L. Complete resolution of all sites of extramedullary disease is required for CR. (CRi): Peripheral blood and marrow results as for CR, but with incomplete recover of counts (platelets < 100 x 10^9/L; neutrophils < 1 x 10^9/L).
Time Frame: Within 3 cycles of treatment initiation
Population: Of the four participants registered on study, three participants were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Treatment (Tagraxofusp, Chemotherapy)
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Participants With a Complete Response
Description: Complete Remission (CR): Normalization of the peripheral blood and bone marrow with 5% or less blasts in normocellular or hypercellular marrow with a granulocyte count of 1 x 10^9/L or above, and platelet count of 100 x 10^9/L. Complete resolution of all sites of extramedullary disease is required for CR.
Time Frame: Within 3 cycles of treatment initiation
Population: Of the four participants registered on study, three participants were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Treatment (Tagraxofusp, Chemotherapy)
Number analyzed (Participants) | 3
Participants | 0

3. Secondary Outcome: Relapsed-free Survival (RFS)
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to two years, 5 months, and 4 days
Population: Of the four participants registered on study, three participants were evaluable for response.
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Tagraxofusp, Chemotherapy)
Number analyzed (Participants) | 3
Months | NA [NA to NA] — There were zero responses in the three evaluable patients.

4. Secondary Outcome: Overall Survival
Description: Kaplan-Meier method will be used to estimate the overall survival.
Time Frame: Up to two years, 5 months, and 4 days
Population: Of the four participants registered on study, three participants were evaluable for response.
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Tagraxofusp, Chemotherapy)
Number analyzed (Participants) | 3
Months | 3.8 [1.7 to 5.3]

ADVERSE EVENTS:
Time Frame: Up to two years, 5 months, and 4 days
Arm/Group | Phase I Treatment (Tagraxofusp, Chemotherapy)
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 4/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Treatment (Tagraxofusp, Chemotherapy) (N=4)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (4)
Non-cardiac chest pain (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Treatment (Tagraxofusp, Chemotherapy) (N=4)
Alanine aminotransferase increased (Investigations) | 4 (7)
Alkaline phosphatase increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Bacteremia (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 1 (2)
Blurred vision (Eye disorders) | 1 (1)
Capillary leak syndrome (Vascular disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Creatinine increased (Investigations) | 2 (3)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Edema limbs (General disorders) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 2 (4)
Fibrinogen decreased (Investigations) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Headache (Nervous system disorders) | 1 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (2)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (5)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 (3)
Hypertension (Vascular disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (6)
INR increased (Investigations) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Investigations - Other, specify (Investigations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (3)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (4)
Somnolence (Nervous system disorders) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT05032183/Prot_SAP_001.pdf